CLINICAL TRIAL: NCT05380739
Title: Working Memory Training and Neural Plasticity in Mild Cognitive Impairment
Brief Title: Memory Training and Neural Plasticity
Acronym: WMTrain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of funding
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexandru Iordan, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00199574
Record Dates: First submitted 2022-04-27; First posted 2022-05-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Working Memory; Training; fMRI
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants in the MCI group will be assigned to receive either in-person (Arm1) or online WM training (Arm2), based on their preference and availability of equipment ensuring a stable internet connection, for 10 training sessions. Participants in the HC group will receive online training (Arm3). Data for HC who received in-person training was already collected (HUM00033133). WM performance in conjunction with brain imaging will be assessed within-subject, twice pre-training (Time1 and Time2) and once post-training (Time3), as well as ~1 month after training (Follow-up). The Time1 vs. Time2 comparison will reveal task-exposure effects, whereas the Time2 vs. Time3 comparison will reveal training effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-Person, MCI (Active Comparator): Participants diagnosed with MCI will undergo 10 sessions of WM training in person.
  Interventions: Behavioral: Working Memory Training
- Online, MCI (Active Comparator): Participants diagnosed with MCI will undergo 10 sessions of WM training online.
  Interventions: Behavioral: Working Memory Training
- Online, Healthy (Active Comparator): Cognitively intact older adults will undergo 10 sessions of WM training online.
  Interventions: Behavioral: Working Memory Training

INTERVENTIONS:
Behavioral: Working Memory Training — A 10-session working memory (WM) training program

SUMMARY:
This study will evaluate the efficacy of working memory training in older adults with amnestic mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Working memory (WM) is the ability to hold information actively in mind and is fundamental for higher-order cognition. This pilot study aims to (1) evaluate the efficacy of WM training in older adults with MCI and (2) understand if and how it works. The study will use behavioral and brain imaging assessments to see whether WM training changes how participants learn and remember information. Functional magnetic resonance imaging (fMRI) and functional near infrared spectroscopy (fNIRS) methods will be used. The study will also use cognitive tests and questionnaires to determine whether participants' cognitive abilities change with training. The study will enroll participants with a diagnosis of MCI as well as cognitively intact older adults (healthy controls, HC).

ELIGIBILITY:
Inclusion Criteria:

* MCI Diagnosis
* Right-handedness
* MRI-eligibility for MRI participants

Exclusion Criteria:

* History of other contributing neurological or medical conditions known to affect cognitive functioning
* Significant mental illness
* Sensory impairments that limit ability to participate
* History of alcohol or drug abuse/dependence

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Gains in WM training task performance | 2 weeks
  Analyses of WM performance for each training session indexed as the mean set-size achieved during each training session for each participant
Changes in brain activation within the WM network | 2 weeks
  Univariate analyses via fMRI and fNIRS, respectively, using units of brain activation (i.e., contrast estimates)

SECONDARY OUTCOMES:
Changes in criterion (fMRI) WM task performance | 2 weeks
  Analyses of WM performance indexed as percent accuracy
Changes in functional connectivity within and between canonical brain networks | 2 weeks
  Graph theory analysis via fMRI and fNIRS, respectively, using measures of connectivity strength (i.e., correlation coefficients)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Iordan, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No